CLINICAL TRIAL: NCT00482092
Title: A Phase III, Multicenter, Placebo-controlled, Randomized, Double-blind Study to Evaluate the Safety and Efficacy of PROCHYMAL® (ex Vivo Cultured Adult Human Mesenchymal Stem Cells) Intravenous Infusion for the Induction of Remission in Subjects Experiencing Treatment-refractory Moderate-to-severe Crohn's Disease
Brief Title: Evaluation of PROCHYMAL® Adult Human Stem Cells for Treatment-resistant Moderate-to-severe Crohn's Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mesoblast, Inc. (Industry)
Responsible Party: Sponsor
Organization: Mesoblast, Ltd. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CRD 603; NCT00609232 (obsolete NCT alias)
Record Dates: First submitted 2007-05-30; First posted 2007-06-04 (Estimated); Last update posted 2022-01-13 (Actual); Status verified 2022-01

CONDITIONS: Crohn's Disease
Keywords: Crohn's disease; adult stem cell therapy
MeSH Terms: conditions — Crohn Disease | interventions — remestemcel-l

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): Participants will receive matching placebo administered as intravenous (IV) infusions.
  Interventions: Drug: Placebo
- Prochymal® - Low dose (Active Comparator): Participants will receive a total dose of Prochymal® 600 x 10^6 cells, IV infusion, on four days, once daily.
  Interventions: Drug: Prochymal®
- Prochymal® - High dose (Active Comparator): Participants will receive a total dose of Prochymal® 1200 x 10^6 cells, IV infusion, on four days, once daily.
  Interventions: Drug: Prochymal®

INTERVENTIONS:
Drug: Prochymal® — Prochymal® IV infusion
  Other Names: Adult Human Mesenchymal Stem Cells
  Arms: Prochymal® - High dose; Prochymal® - Low dose
Drug: Placebo — Prochymal® Placebo-matching IV infusion
  Arms: Placebo

SUMMARY:
Protocol 603 is enrolling subjects with moderate-to-severe Crohn's disease who are intolerant to, or have previously failed therapy with, at least one steroid and at least one immunosuppressant and a biologic monoclonal anti-body to tumor necrosis factor alpha. The protocol investigates the safety and efficacy of using PROCHYMAL® adult human stem cells to induce remission. PROCHYMAL is delivered through a vein in the arm four times over two weeks, for approximately an hour each time.

DETAILED DESCRIPTION:
A significant number of individuals with Crohn's disease do not find relief with existing steroidal, immunosuppressive, or biologic therapies, and are forced to seek surgery or other drastic measures for treatment.

PROCHYMAL® adult human stem cells are manufactured from healthy, volunteer donors, extensively tested, and are stored to be available as needed. Human and animal studies have shown that the cells do not require any donor-recipient matching. The cells may have both immunosuppressive and healing benefits in Crohn's disease. The cells naturally migrate specifically to sites of inflammation, so their effects are believed to be local and self-limiting rather than systemic.

Protocol 603 is enrolling subjects to evaluate the ability of PROCHYMAL to induce remission in subjects with moderate-to-severe disease (Crohn's disease activity index -- CDAI -- of between 250 and 450, inclusive) who have failed or been intolerant of at least one drug in each of the steroid, immunosuppressant, and biologic classes.

ELIGIBILITY:
Inclusion Criteria:

* failed (within last 2 yr) or intolerant of at least one steroid AND at least one immunosuppressant AND at EXACTLY one biologic
* CDAI between 250 and 450, inclusive
* endoscopically or radiographically confirmed Crohn's disease of ileus or colon or both
* C-Reactive Protein Test (CRP) of at least 5 mg/l (0.5 mg/dl)*OR* CDAI of at least 300
* weight between 40 and 150 kg, inclusive
* adequate renal function
* negative tuberculosis skin (PPD) test (or evaluated low risk of TB activation)

Exclusion Criteria:

* HIV or hepatitis infection active
* allergy to CT contrast agents, or to bovine or porcine products
* symptomatic fibrostenotic Crohn's disease
* permanent ostomy
* biologic therapy within past 90 d
* prednisone greater than 20 mg/d within past month
* short-bowel syndrome
* total parenteral nutrition
* abnormal liver function
* malignancy active within past 5 years (except completely resected basal or squamous cell carcinoma of skin)
* enteric pathogens, including C. difficile
* history of colonic mucosal dysplasia
* current or prior evidence of tuberculosis (TB) (unless risk of activation or re-activation deemed low)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 330 (Actual)
Dates: Start 2007-09-17 (Actual); Primary Completion 2014-09-15 (Actual); Study Completion 2014-09-15 (Actual)

PRIMARY OUTCOMES:
Disease remission (CDAI at or below 150) | 28 days

SECONDARY OUTCOMES:
Disease improvement (Reduction by at least 100 points in CDAI) | 28 days
Improvement in quality of life (IBDQ) | 28 days
Reduction in number of draining fistulas | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Mahboob Rahman, MD, Study Director — Mesoblast, Inc.
Locations (56):
- United States (47):
  - University of Southern California University Hospital, Los Angeles, California
  - University of California, San Francisco, San Francisco, California
  - Western States Clinical Research, Wheat Ridge, Colorado
  - Clinical Research of West Florida, Clearwater, Florida
  - Borland-Groover Clinic, Jacksonville, Florida
  - Shafran Gastroenterology Center, Winter Park, Florida
  - Atlanta Gastroenterology Associates, Atlanta, Georgia
  - University of Chicago Medical Center, Chicago, Illinois
  - Carle Clinic Association, Urbana, Illinois
  - Indiana University Medical Center, Indianapolis, Indiana
  - Cotton-O'Neil Clinical Research Center, Topeka, Kansas
  - University of Kentucky Hospital, Lexington, Kentucky
  - University of Louisville Hospital, Louisville, Kentucky
  - Gulf Coast Research, Baton Rouge, Louisiana
  - University of Maryland, Baltimore, Baltimore, Maryland
  - National Institutes of Health, Bethesda, Maryland
  - Chevy Chase Clinical Research, Chevy Chase, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Womens Hospital, Boston, Massachusetts
  - Clinical Pharmacology Study Group, Worcester, Massachusetts
  - Center for Clinical Studies, Dearborn, Michigan
  - Center for Digestive Health, Troy, Michigan
  - University of Minnesota Hospital, Minneapolis, Minnesota
  - St Louis Center for Clinical Studies, St Louis, Missouri
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Weill Cornell Medical College, New York, New York
  - Mount Sinai School of Medicine, New York, New York
  - Rochester Institute for Digestive Diseases, Rochester, New York
  - Rochester General Hospital, Rochester, New York
  - University Hospital and Medical Center, Stony Brook, New York
  - Charlotte Gastroenterology and Hepatology, Charlotte, North Carolina
  - Pinehurst Medical Clinic, Pinehurst, North Carolina
  - Wake Forest University, Winston-Salem, North Carolina
  - Gastroenterology United of Tulsa, Tulsa, Oklahoma
  - Options Health Research, Tulsa, Oklahoma
  - Allegheney Center for Digestive Health, Pittsburgh, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Gastroenterology Center of the Midsouth, Germantown, Tennessee
  - Nashville GI Specialists, Nashville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Baylor University Medical Center, Dallas, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - University of Texas Health Science Center, Houston, Texas
  - University of Vermont, Burlington, Vermont
  - Digestive and Liver Disease Specialists, Norfolk, Virginia
  - McGuire Research Institute, Richmond, Virginia
  - Seattle Gastroenterology Associates, Seattle, Washington
- Australia (2):
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Royal Melbourne Hospital, Melbourne, Victoria
- Canada (5):
  - University of Calgary, Calgary, Alberta
  - University of Alberta Hospital, Edmonton, Alberta
  - Health Science Centre, Winnipeg, Manitoba
  - London Health Sciences Centre, London, Ontario
  - Mount Sinai Hospital, Toronto, Ontario
- New Zealand (2):
  - University of Otago, Christchurch
  - Waikato Hospital, Hamilton